CLINICAL TRIAL: NCT07336121
Title: Assessment of Outcome and Tolerability of High Velocity Nasal Insufflation and Continuous Positive Airway Pressure in Children With Acute Respiratory Distress
Brief Title: HVNI vs CPAP in Children With Acute Respiratory Distress
Acronym: P-HVNI-CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MD 11/2023; FMASU MD 11 /2023 (Other: Research Ethics Committee-Faculty of Medicine-ASU)
Record Dates: First submitted 2025-12-14; First posted 2026-01-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2023-01

CONDITIONS: Community Acquired Pneumonia; Bronchiolitis
Keywords: High -Velocity Nasal Insufflation; Continuous positive Airway Pressure; Pediatric Acute Respiratory Distress; pediatric intensive care unit
MeSH Terms: conditions — Community-Acquired Pneumonia; Bronchiolitis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Velocity Nasal Insufflation (HVNI) (Active Comparator): Children aged 1 month to 5 years with acute respiratory distress admitted to the PICU will receive respiratory support using High Velocity Nasal Insufflation after failure of low-flow oxygen therapy. Outcomes and tolerability will be assessed clinically and by daily lung ultrasound score during PICU stay.
  Interventions: Device: High Velocity Nasal Insufflation (HVNI)
- Nasal Continuous Positive Airway Pressure (Nasal CPAP) (Active Comparator): Children aged 1 month to 5 years with acute respiratory distress admitted to the PICU will receive respiratory support using nasal Continuous Positive Airway Pressure after failure of low-flow oxygen therapy. Outcomes and tolerability will be assessed clinically and by daily lung ultrasound score during PICU stay.
  Interventions: Device: Nasal Continuous Positive Airway Pressure (Nasal CPAP)

INTERVENTIONS:
Device: High Velocity Nasal Insufflation (HVNI) — High Velocity Nasal Insufflation will be delivered using a heated, humidified nasal cannula system to children aged 1 month to 5 years with acute respiratory distress who failed low-flow oxygen therapy. Therapy will be initiated and adjusted according to clinical condition and institutional PICU protocol. Patients will be monitored clinically and by daily lung ultrasound score during PICU stay.
  Arms: High Velocity Nasal Insufflation (HVNI)
Device: Nasal Continuous Positive Airway Pressure (Nasal CPAP) — Nasal Continuous Positive Airway Pressure will be delivered via nasal interface providing continuous positive airway pressure with supplemental oxygen to children aged 1 month to 5 years with acute respiratory distress who failed low-flow oxygen therapy. Settings will be adjusted according to clinical response and institutional PICU protocol. Patients will be monitored clinically and by daily lung ultrasound score during PICU stay.
  Arms: Nasal Continuous Positive Airway Pressure (Nasal CPAP)

SUMMARY:
Acute breathing problems are a common reason for children to be admitted to the pediatric intensive care unit, and many of these children need breathing support without a breathing tube. High-Velocity Nasal Insufflation (HVNI) and nasal Continuous Positive Airway Pressure (nCPAP) are commonly used to help children breathe, but there is limited information comparing how well they work and how comfortable they are for children. This study aims to compare the clinical outcomes and tolerability of HVNI and nCPAP in children aged 1 month to 5 years with acute respiratory distress admitted to the pediatric intensive care unit, using clinical assessment and lung ultrasound findings.

DETAILED DESCRIPTION:
Acute respiratory distress represents a major cause of morbidity and mortality in infants and young children and accounts for a significant proportion of pediatric intensive care unit admissions. A considerable number of affected children fail conventional low-flow oxygen therapy and require escalation to non-invasive respiratory support.

High Velocity Nasal Insufflation delivers heated and humidified oxygen at high flow rates through nasal cannulae and may improve oxygenation by washing out nasopharyngeal dead space, reducing inspiratory resistance, and providing a degree of positive end-expiratory pressure. Nasal Continuous Positive Airway Pressure delivers a continuous distending airway pressure with supplemental oxygen, improving lung recruitment, reducing atelectasis, and enhancing ventilation-perfusion matching.

Both modalities are commonly used in pediatric intensive care practice; however, evidence comparing their clinical effectiveness, tolerability, and impact on lung aeration in young children remains inconclusive. Lung ultrasound has emerged as a reliable, non-invasive bedside tool for assessment of lung aeration and disease severity in critically ill children.

This prospective interventional study will enroll 80 children aged 1 month to 5 years admitted to the pediatric intensive care unit with acute respiratory distress who have failed low-flow oxygen therapy. Patients will be randomized into two groups: one group receiving High Velocity Nasal Insufflation and the other receiving nasal Continuous Positive Airway Pressure. All patients will undergo daily clinical assessment and lung ultrasound scoring during their pediatric intensive care unit (PICU) stay. Tolerability will be evaluated using the FLACC (Face, Legs, Activity, Cry, Consolability) pain scale.

The primary outcome is improvement in lung aeration as assessed by lung ultrasound score. Secondary outcomes include assessment of clinical response to therapy based on respiratory rate, oxygen saturation (SpO₂), and need for escalation of respiratory support . The results of this study aim to provide evidence to guide selection of optimal non-invasive respiratory support in children with acute respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 5 years
* Admitted to the Pediatric Intensive Care Unit (PICU)
* Diagnosed with acute respiratory distress
* Failure of low-flow nasal oxygen therapy
* Requiring non-invasive respiratory support
* Informed consent obtained from parent or legal guardian

Exclusion Criteria:

* Presence of congenital or acquired cardiac disease
* Neuromuscular disorders
* Chronic lung disease
* History of recurrent wheezing
* History of cardio-respiratory arrest
* Presence of significant comorbid chronic illness
* Contraindication to non-invasive ventilation

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement in lung aeration assessed by lung ultrasound score | At Baseline, pre procedural , 48 hours .
  To compare the effectiveness of High Velocity Nasal Insufflation versus Nasal Continuous Positive Airway Pressure in improving lung aeration in children with acute respiratory distress, assessed by daily lung ultrasound score during PICU stay.
  The LUS ranges from 0 to 36, where higher scores indicate worse lung aeration and lower scores indicate improvement.

SECONDARY OUTCOMES:
Clinical improvement of respiratory distress assessed by Modified Respiratory Distress Score | Baseline and 48 hours after initiation of respiratory support
  Clinical improvement assessed using a Modified Respiratory Distress Score(MRDS), which incorporates respiratory rate (breaths/min), oxygen saturation measured by pulse oximetry (SpO₂, %), and fraction of inspired oxygen (FiO₂, %).
  The MRDS ranges from 0 to 12, where higher scores indicate more severe respiratory distress and lower scores indicate clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek A. Abdelgawad, MD, Principal Investigator — Ain Shams University
Locations (1):
- Pediatric Intensive Care Units, Children Hospital, Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Result] Liu C, Cheng WY, Li JS, Tang T, Tan PL, Yang L. High-Flow Nasal Cannula vs. Continuous Positive Airway Pressure Therapy for the Treatment of Children <2 Years With Mild to Moderate Respiratory Failure Due to Pneumonia. Front Pediatr. 2020 Nov 13;8:590906. doi: 10.3389/fped.2020.590906. eCollection 2020. PMID 33304868
- See also: High flow nasal cannula therapy versus continuous positive airway pressure and nasal positive pressure ventilation in infants with severe bronchiolitis: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/34909101/

DOCUMENTS (2):
  • Study Protocol (2023-01-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT07336121/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT07336121/SAP_001.pdf